CLINICAL TRIAL: NCT01896999
Title: A Phase I Study With an Expansion Cohort/Randomized Phase II Study of the Combinations of Ipilimumab, Nivolumab and Brentuximab Vedotin in Patients With Relapsed/Refractory Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin and Nivolumab With or Without Ipilimumab in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01275; NCI-2013-01275 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E4412; S14-00011; E4412 (Other: ECOG-ACRIN Cancer Research Group); E4412 (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Classic Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Brentuximab Vedotin; Ipilimumab; CTLA-4 Antigen; Nivolumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase I Arm I (brentuximab vedotin, ipilimumab) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on day 1 of cycles 1-16 and ipilimumab IV over 90 minutes on day 1 of cycles 1-4, 8, 12, and 16. Treatment repeats every 21 days for up to 16 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or PET scan throughout the trial. Patients undergo blood sample collection and may undergo tumor biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Positron Emission Tomography
- Phase I Arm II (brentuximab vedotin, nivolumab) (Experimental): Patients receive brentuximab vedotin IV over 90 minutes on day 1 of cycles 1-16 and nivolumab IV over 30 minutes on day 1 of cycles 1-46. Treatment repeats every 21 days for up to 16 cycles and every 14 days beginning cycle 17 for up to 46 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or PET scan throughout the trial. Patients undergo blood sample collection and may undergo tumor biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Biological: Nivolumab; Procedure: Positron Emission Tomography
- Phase I Arm III (brentuximab vedotin, nivolumab, ipilimumab) (Experimental): Patients receive brentuximab vedotin IV over 90 minutes on day 1 of cycles 1-16, nivolumab IV over 30 minutes on day 1 of cycles 1-46, and ipilimumab IV over 30 minutes on day 1 every 12 weeks for up to 9 doses. Treatment repeats every 21 days for up to 16 cycles and every 14 days beginning cycle 17 for up to 46 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or PET scan throughout the trial. Patients undergo blood sample collection and may undergo tumor biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Biological: Ipilimumab; Biological: Nivolumab; Procedure: Positron Emission Tomography
- Phase II Arm I (brentuximab vedotin, nivolumab) (Experimental): Patients receive brentuximab vedotin IV over 90 minutes on day 1 of cycles 1-16 and nivolumab IV over 30 minutes on day 1 of cycles 1-34. Treatment repeats every 21 days for up to 34 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or PET scan throughout the trial. Patients undergo blood sample collection and may undergo tumor biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Biological: Nivolumab; Procedure: Positron Emission Tomography
- Phase II Arm II (brentuximab vedotin, nivolumab, ipilimumab) (Experimental): Patients receive brentuximab vedotin IV over 90 minutes on day 1 of cycles 1-16, nivolumab IV over 30 minutes on day 1 of cycles 1-34, and ipilimumab IV over 30 minutes on day 1 every 12 weeks for up to 9 doses. Treatment repeats every 21 days for up to 34 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or PET scan throughout the trial. Patients undergo blood sample collection and may undergo tumor biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Biological: Ipilimumab; Biological: Nivolumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN 35; SGN-35; SGN35
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Phase I Arm I (brentuximab vedotin, ipilimumab); Phase I Arm III (brentuximab vedotin, nivolumab, ipilimumab); Phase II Arm II (brentuximab vedotin, nivolumab, ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Phase I Arm II (brentuximab vedotin, nivolumab); Phase I Arm III (brentuximab vedotin, nivolumab, ipilimumab); Phase II Arm I (brentuximab vedotin, nivolumab); Phase II Arm II (brentuximab vedotin, nivolumab, ipilimumab)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I/II trial studies the side effects and best dose of ipilimumab and nivolumab when given together with brentuximab vedotin, and how well they work in treating patients with Hodgkin lymphoma that has returned after a period of improvement (recurrent) or has not responded to previous treatment (refractory). Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Brentuximab vedotin is a monoclonal antibody, brentuximab, linked to a toxic agent called vedotin. Brentuximab attaches to CD30 positive cancer cells in a targeted way and delivers vedotin to kill them. It is not known whether giving brentuximab vedotin and nivolumab with or without ipilimumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of the combinations of brentuximab vedotin and ipilimumab, brentuximab vedotin and nivolumab, and brentuximab vedotin, ipilimumab, and nivolumab. (Phase I) II. To evaluate the complete response (CR) rate for the regimens of brentuximab vedotin and nivolumab compared to brentuximab vedotin, ipilimumab, and nivolumab. (Phase II; adult cohort [aged >= 18 years]) III. To characterize the safety and toxicity of treatment combination in the pediatric population. (Phase II; pediatric cohort [aged 12-17 years])

SECONDARY OBJECTIVES:

I. To evaluate complete response (CR) rate, partial response (PR) rate and overall response rate (ORR), for the combinations of brentuximab vedotin and ipilimumab, brentuximab vedotin and nivolumab, and brentuximab vedotin, ipilimumab, and nivolumab. (Phase I) II. To evaluate the duration of remission (DOR) to these combinations and compare with the DOR achieved with the most recent prior systemic therapy. (Phase I) III. To evaluate the progression-free survival (PFS) and the overall survival (OS) in patients receiving the combination of brentuximab vedotin and ipilimumab, brentuximab vedotin and nivolumab, and brentuximab vedotin, ipilimumab, and nivolumab. (Phase I) IV. To evaluate the ORR, PR, and stable disease (SD) rate for the combinations of brentuximab vedotin and nivolumab and brentuximab vedotin, ipilimumab, and nivolumab. (Phase II) V. To evaluate the DOR to these combinations and compare with the DOR achieved with the most recent prior systemic therapy. (Phase II) VI. To evaluate the 5 year PFS and OS in patients receiving the combinations of brentuximab vedotin and nivolumab and brentuximab vedotin, ipilimumab, and nivolumab. (Phase II) VII. To further evaluate the safety and characterize the toxicity for the combinations of brentuximab vedotin and nivolumab, and brentuximab vedotin, ipilimumab, and nivolumab. (Phase II)

CORRELATIVE STUDY OBJECTIVES:

I. To evaluate the ability of these combinations to alter tumor specific T cell immunity. (Phase I) II. To evaluate the effects of these combinations on systemic immunity. (Phase I) III. To evaluate a panel of cytokine and T cell specific biomarkers from the peripheral blood as a potential immune signature of treatment response to therapy with these combinations for patients with relapsed/refractory Hodgkin lymphoma (HL). (Phase I) IV. To evaluate using gene expression profiling (GEP) a signature of response to these novel combinations of an antibody drug conjugate with immunomodulatory therapy. (Phase I) V. To evaluate the ability of these combinations to alter tumor specific T cell immunity, and circulating T cell phenotypes, in patients as a function of treatment response at multiple timepoints during therapy. (Phase II) VI. To evaluate peripheral blood cytokine profiles in responding and resistant patients at multiple timepoints during therapy. (Phase II) VII. To evaluate using GEP a signature of response versus (vs.) resistance to these novel combinations of an antibody drug conjugate with immunomodulatory therapy. (Phase II) VIII. To evaluate the influence of human gut microbiome dysbiosis on HL lymphomagenesis and the systemic immune response. (Phase II)

IMAGING CORRELATIVE STUDY OBJECTIVES:

I. To evaluate atypical response patterns with currently available response evaluation criteria. (Phase II) II. To correlate response evaluated using currently available response evaluation criteria with duration of response (PFS, event free survival [EFS], failure free survival [FFS]). (Phase II) III. To evaluate response patterns in different immunotherapy treatment schemes and correlate with historical data using chemotherapy. (Phase II) IV. To correlate imaging changes in all treatment schemes quantitatively with PFS. (Phase II)

EXPLORATORY OBJECTIVES:

I. Evaluate outcomes (CR, PFS) between patients with/without prior transplants. (Phase II) II. Evaluate outcomes (PFS, OS) between the patients who stay on treatment and do not go to transplant in both arms (the post auto and the few others who don't want transplant) vs the patients who go off for transplant. (Phase II) III. Evaluate outcomes (CR, PFS) in pediatric population (age 12 to < 18 years of age) vs. adult population. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of brentuximab vedotin, ipilimumab, and nivolumab followed by a phase II study.

PHASE I: Patients are assigned into 1 of 3 arms.

ARM I: Patients receive brentuximab vedotin intravenously (IV) over 90 minutes on day 1 of cycles 1-16 and ipilimumab IV over 30 minutes on day 1 of cycles 1-4, 8, 12, and 16. Treatment repeats every 21 days for up to 16 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive brentuximab vedotin IV over 90 minutes on day 1 of cycles 1-16 and nivolumab IV over 30 minutes on day 1 of cycles 1-46. Treatment repeats every 21 days for up to 16 cycles and every 14 days beginning cycle 17 for up to 46 cycles in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive brentuximab vedotin IV over 90 minutes on day 1 of cycles 1-16, nivolumab IV over 30 minutes on day 1 of cycles 1-46, and ipilimumab IV over 30 minutes on day 1 every 12 weeks for up to 9 doses. Treatment repeats every 21 days for up to 16 cycles and every 14 days beginning cycle 17 for up to 46 cycles in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive brentuximab vedotin IV over 30 minutes on day 1 of cycles 1-16 and nivolumab IV over 90 minutes on day 1 of cycles 1-34. Treatment repeats every 21 days for up to 34 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive brentuximab vedotin IV over 90 minutes on day 1 of cycles 1-16, nivolumab IV over 30 minutes on day 1 of cycles 1-34, and ipilimumab IV over 30 minutes on day 1 every 12 weeks for up to 9 doses. Treatment repeats every 21 days for up to 34 cycles in the absence of disease progression or unacceptable toxicity.

All patients also undergo computed tomography (CT) or positron emission tomography (PET) scan throughout the trial. Patients undergo blood sample collection and may undergo tumor biopsy on study.

After completion of phase I study treatment, patients are followed up every 3 months for 1 year, then every 6 months for 2 years. After completion of phase II study treatment, patients are followed up for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I (ARMS A, B, C, D, E, F, G, H, I, X, Y, Z)
* Age >= 18 years
* Patients must have pathologically confirmed relapsed or refractory classical Hodgkin lymphoma (cHL); a biopsy at any relapse is acceptable; other histologies including lymphocyte predominant (LP) HL are not permitted
* Patients must have relapsed after first line chemotherapy; may have relapsed after autologous or allogeneic stem cell transplant, or have primary refractory disease; no upper limit for number of prior therapies; if status post allogeneic stem cell transplant, no active graft versus host disease
* Patients may have received prior brentuximab vedotin, but must not have received brentuximab vedotin within 6 months prior to registration, and must not have relapsed within 6 months of receiving previous brentuximab vedotin; patients may not have received prior nivolumab or PD1/PDL1 axis agents; patients in the nivolumab/brentuximab cohorts ONLY (D, E, F, Y) may have received prior ipilimumab
* Patients may have received other prior activating immunotherapies (i.e. checkpoint inhibitors), but must not have received them within 6 months prior to registration, and there must be no serious unresolved complication of therapy at the time of registration; for the purposes of this study monoclonal antibodies and antibody drug conjugates are not considered to be activating immunotherapies and there are no additional time restrictions on prior exposure to these agents (except prior brentuximab vedotin)
* Eastern Cooperative Oncology Group (ECOG)-American College of Radiology Imaging Network (ACRIN) performance status between 0-2
* Patients must have measurable disease; baseline measurements and evaluations must be obtained within 4 weeks of registration to the study; abnormal PET scans will not constitute evaluable disease unless verified by a diagnostic quality CT scan; patients must use the same imaging modality (CT or PET/CT) throughout the study
* Patient must not be pregnant or breast-feeding due to risk of fetal harm by the chemotherapeutic agents prescribed in this protocol; all patients of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; a patient of childbearing potential is anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient of childbearing potential and/or sexually active patients must either abstain from sexual intercourse for the duration of their participation in the study or agree to use both single barrier contraception and birth control pills or implants for at least one week prior to the start of the study drug and continuing for 5 months after the last dose of study drug (for patients of childbearing potential) and for 7 months after the last dose of study drug (for patients who are sexually active with anyone of childbearing potential); should a patient become pregnant or suspect pregnancy while the patient or their partner is participating in this study, the patient (or the participating partner) should inform the treating physician immediately
* Patients must have no evidence of dyspnea at rest and a pulse oximetry > 92% while breathing room air
* Patients must have forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) > 60% by pulmonary function test (PFT), unless due to large mediastinal mass from HL; carbon monoxide diffusion capacity (DLCO), FEV1, and FVC all > 50% predicted value; all pulmonary function tests must be obtained within one month prior to registration
* Absolute neutrophil count (ANC) >= 1500/mcL (1.5 x 10^9/L) (obtained within 2 weeks prior to registration)
* Platelets >= 75,000/mcL (75 x 10^9/L) (obtained within 2 weeks prior to registration)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) (obtained within 2 weeks prior to registration)
* Bilirubin =< 2 x upper limit of normal (ULN) (unless documented Gilbert's syndrome, for which bilirubin =< 3 x upper limit of normal [ULN] is permitted) (obtained within 2 weeks prior to registration)
* Calculated creatinine clearance by Cockcroft-Gault formula >= 30 ml/min (obtained within 2 weeks prior to registration)
* No evidence of prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical carcinoma or any surgically- or radiation-cured malignancy continuously disease free for >= 5 years so as not to interfere with interpretation of radiographic response
* Patient must have no current or prior history of central nervous system (CNS) involvement
* All prior therapy must have been completed at least 21 days prior to enrollment; no concomitant anti lymphoma therapy, including systemic corticosteroids for the purpose of treatment of lymphoma are allowed; topical steroids are allowed
* No history of Steven's Johnson's syndrome, toxic epidermal necrolysis (TEN)s syndrome, or motor neuropathy
* Human immunodeficiency virus (HIV) positive patients are allowed on this study if they have a CD4 count > 400, and are on a stable antiviral regimen; patients with poorly controlled HIV or other chronic active viral infections will be excluded
* Patients must not have autoimmune disorders or conditions of immunosuppression that require current ongoing treatment with systemic corticosteroids (or other systemic immunosuppressants), including oral steroids (i.e., prednisone, dexamethasone) or continuous use of topical steroid creams or ointments or ophthalmologic steroids; a history of occasional (but not continuous) use of steroid inhalers is allowed

  * Replacement doses of steroids for patients with adrenal insufficiency are allowed; patients who discontinue use of these classes of medication for at least 2 weeks prior to initiation of study treatment are eligible if, in the judgment of the treating physician investigator, the patient is not likely to require resumption of treatment with these classes of drugs during the study
  * Exclusion from this study also includes patients with a history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjogren's syndrome, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and Myasthenia Gravis); other CNS autoimmune disease (e.g., Multiple sclerosis); patients with autoimmune hypothyroid disease or type I diabetes on replacement treatment are eligible
* Patients must not have grade 2 or greater peripheral sensory neuropathy
* Patients must not have New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia
* Patients must not have previously existing hypersensitivity to brentuximab vedotin or ipilimumab
* Patients must not have a serious medical or psychiatric illness likely to interfere with study participation
* Patients must not be participating in any other clinical trial or taking any other experimental medications within 21 days prior to registration
* Routine vaccinations, including seasonal influenza, should be given at least 2 weeks prior to study treatment; vaccines are not prohibited on study, but must be given at least 6 weeks after cycle 1 and not within 7 days of treatment
* Patients registering to Arms D, E, F, G, H, I, X, Y must not currently be smoking tobacco or other substances and must not have smoked within the past 6 months
* RANDOMIZED PHASE II (ARMS K AND L): Age >= 12 years

  * Pediatric patients will include any patients < 18 years of age
* RANDOMIZED PHASE II (ARMS K AND L): Patients must have pathologically confirmed relapsed or refractory classical Hodgkin lymphoma (cHL); a biopsy at any relapse is acceptable; other histologies including lymphocyte predominant (LP) HL are not permitted
* RANDOMIZED PHASE II (ARMS K AND L): Patients must have relapsed after first line chemotherapy; may have relapsed after autologous stem cell transplant, or have primary refractory disease; no upper limit for number of prior therapies; patient must not have received a prior allogeneic stem cell transplant (out of risk of reactivation of pulmonary graft versus host disease [GVHD])
* RANDOMIZED PHASE II (ARMS K AND L): Patients may have received prior brentuximab vedotin, but must not have received brentuximab vedotin within 6 months prior to registration, and must not have relapsed within 6 months of receiving previous brentuximab vedotin; patients may not have received prior nivolumab or PD1/PDL1 axis agents; patients may not have received prior ipilimumab
* RANDOMIZED PHASE II (ARMS K AND L): Patients may not have received other prior activating immunotherapies (i.e. checkpoint inhibitor therapies); for the purposes of this study monoclonal antibodies and antibody drug conjugates are not considered to be activating immunotherapies and there are no additional time restrictions on prior exposure to these agents (except prior brentuximab vedotin)
* RANDOMIZED PHASE II (ARMS K AND L): Adult patient (>= 18 years of age) ECOG-ACRIN performance status between 0-2

  * Pediatric patients (16-17 years of age) must have a Karnofsky performance level >= 50%
  * Pediatric patients (12-15 years of age) must have a Lansky performance level >= 50
* RANDOMIZED PHASE II (ARMS K AND L): Patients must have measurable disease; baseline measurements and evaluations must be obtained within 4 weeks of registration to the study; abnormal PET scans will not constitute evaluable disease unless verified by a diagnostic quality CT scan; patients must use the same imaging modality (CT or PET/CT) throughout the study
* RANDOMIZED PHASE II (ARMS K AND L): Patient must not be pregnant or breast-feeding due to risk of fetal harm by the chemotherapeutic agents prescribed in this protocol; all patients of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; a patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* RANDOMIZED PHASE II (ARMS K AND L): Patient of childbearing potential and/or sexually active patient must either abstain from sexual intercourse for the duration of their participation in the study or agree to use both double barrier contraception and birth control pills or implants for at least one week prior to the start of the study drug and continuing for 5 months after the last dose of study drug (for patients of childbearing potential) and for 7 months after the last dose of study drug (for patients who are sexually active with anyone of childbearing potential); should a patient become pregnant or suspect pregnancy while the patient or their partner is participating in this study, the patient (or the participating partner) should inform the treating physician immediately
* RANDOMIZED PHASE II (ARMS K AND L): Patients with impaired decision-making capacity are eligible with legally authorized representative
* RANDOMIZED PHASE II (ARMS K AND L): Patients must have no evidence of dyspnea at rest and a pulse oximetry > 92% while breathing room air
* RANDOMIZED PHASE II (ARMS K AND L): Patients must have FEV1/FVC > 60% by pulmonary function test (PFT), unless due to large mediastinal mass from HL; carbon monoxide diffusion capacity (DLCO), FEV1, and FVC all > 50% predicted value; all pulmonary function tests must be obtained within one month prior to registration
* RANDOMIZED PHASE II (ARMS K AND L): ANC >= 1500/mcL (1.5 x 0^9/L) (obtained within 2 weeks prior to registration)
* RANDOMIZED PHASE II (ARMS K AND L): Platelets >= 75,000/mcL (75 x 10^9/L) (obtained within 2 weeks prior to registration)
* RANDOMIZED PHASE II (ARMS K AND L): AST/ALT =< 2.5 x upper limit of normal (ULN) for age (obtained within 2 weeks prior to registration)
* RANDOMIZED PHASE II (ARMS K AND L): Bilirubin =< 2 x upper limit of normal (ULN) (unless documented Gilbert's syndrome, for which bilirubin =< 3 x upper limit of normal [ULN] is permitted) (obtained within 2 weeks prior to registration)
* RANDOMIZED PHASE II (ARMS K AND L): Adult patients (>= 18 years old) must have a calculated creatinine clearance by Cockcroft-Gault formula >= 30 ml/min (obtained within 2 weeks prior to registration)
* RANDOMIZED PHASE II (ARMS K AND L): Pediatric patients (< 18 years old) must have a creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or serum creatinine based on age/gender as follows:

  * Age: maximum serum creatinine (mg/dL)

    * < 13 years: male (1.2), female (1.2)
    * 13 to < 16 years: male (1.5), female (1.4)
    * >= 16 years: male (1.7), female (1.4)
* RANDOMIZED PHASE II (ARMS K AND L): No evidence of prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical carcinoma or any surgically- or radiation-cured malignancy continuously disease free for >= 5 years so as not to interfere with interpretation of radiographic response
* RANDOMIZED PHASE II (ARMS K AND L): Patient must have no current or prior history of CNS involvement
* RANDOMIZED PHASE II (ARMS K AND L): All prior therapy must have been completed at least 21 days prior to enrollment (6 weeks for nitrosoureas or mitomycin C); no concomitant anti lymphoma therapy, including systemic corticosteroids for the purpose of treatment of lymphoma are allowed; topical steroids are allowed
* RANDOMIZED PHASE II (ARMS K AND L): No history of Steven's Johnson's syndrome, TENs syndrome, or motor neuropathy
* RANDOMIZED PHASE II (ARMS K AND L): HIV positive patients are eligible provided they meet the other protocol criteria including the following:

  * Long term survival expected were it not for the cHL
  * HIV viral loads undetectable by standard clinical HIV testing
  * Willing to adhere to effective combination antiretroviral therapy
* RANDOMIZED PHASE II (ARMS K AND L): Patients must not have autoimmune disorders, prior solid organ transplant, or conditions of immunosuppression that require current ongoing treatment with systemic corticosteroids (or other systemic immunosuppressants), including oral steroids (i.e., prednisone, dexamethasone) or continuous use of topical steroid creams or ointments or ophthalmologic steroids; a history of occasional (but not continuous) use of steroid inhalers is allowed; replacement doses of steroids for patients with adrenal insufficiency are allowed; patients who discontinue use of steroid medication for at least 2 weeks prior to initiation of therapy are eligible if, in the judgment of the treating physician investigator, the patient is not likely to require resumption of treatment with these classes of drugs during the study; exclusion from this study also includes patients with a history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjogren's syndrome, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and Myasthenia Gravis); other CNS autoimmune disease (e.g., Multiple sclerosis); patients with autoimmune hypothyroid disease or type I diabetes on replacement treatment are eligible
* RANDOMIZED PHASE II (ARMS K AND L): Patients must not have grade 2 or greater peripheral sensory neuropathy
* RANDOMIZED PHASE II (ARMS K AND L): Patients must not have NYHA class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia
* RANDOMIZED PHASE II (ARMS K AND L): Patients must not have previously existing hypersensitivity to brentuximab vedotin or ipilimumab
* RANDOMIZED PHASE II (ARMS K AND L): Patients must not have a serious medical or psychiatric illness likely to interfere with study participation
* RANDOMIZED PHASE II (ARMS K AND L): Patients must not be participating in any other clinical trial or taking any other experimental medications within 21 days prior to registration
* RANDOMIZED PHASE II (ARMS K AND L): Routine vaccinations, including seasonal influenza, should be given at least 2 weeks prior to study treatment; vaccines are not prohibited on study, but must be given at least 6 weeks after cycle 1 and not within 7 days of treatment
* RANDOMIZED PHASE II (ARMS K AND L): Patients must not currently be smoking tobacco or other agents; vaping is not allowed
* RANDOMIZED PHASE II (ARMS K AND L): Patients must not have a history of or evidence of cardiovascular risks including any of the following:

  * QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec at baseline
  * History of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within the past 24 weeks prior to registration
  * History prior to registration or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Left ventricular ejection fraction (LVEF) =< lower limit of normal on cardiac echocardiogram (echo) or multigated acquisition scan (MUGA)
  * Intra-cardiac defibrillator
  * History of abnormal cardiac valve morphology (>= grade 2) documented by ECHO; (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study); subjects with moderate valvular thickening should not be entered on study
  * History or evidence of current clinically significant uncontrolled cardiac arrhythmias; clarification: subjects with atrial fibrillation controlled for > 30 days prior to dosing are eligible
  * Treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2014-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of each combination (Phase I) | 21 days
  MTD defined as the highest dose level at which less than 33% of 6 patients experience a dose limiting toxicity, will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Upon completion of the trial, frequency of subjects experiencing toxicities will be tabulated. Toxicities will be assessed and graded according to CTCAE version 4.0 terminology. Exact 95% confidence intervals (CI) around the toxicity proportions will be calculated.
CR rate (Phase II) | Up to 10 years
  The analysis of CR between two arms will be performed using exact Cochran-Mantel-Haenszel (CMH) test stratifying on prior brentuximab vedotin (BV) (yes versus [vs.] no) and age (< 18 vs. >= 18). Multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes.

SECONDARY OUTCOMES:
Complete response (CR) rate (Phase I) | Up to 3 years
  Assessed using the Revised Response Criteria for Malignant Lymphoma and reported along with the 95% CI.
Partial response (PR) rate (Phase I) | Up to 3 years
  Assessed using the Revised Response Criteria for Malignant Lymphoma and reported along with the 95% CI.
Overall response rate (ORR) rate (Phase I) | Up to 3 years
  Assessed using the Revised Response Criteria for Malignant Lymphoma and reported along with the 95% CI.
Duration of response (DOR) (Phase I) | From the documented beginning of response up to 3 years
  DOR will be estimated using Kaplan-Meier methodology. Greenwood's formula will be used to calculate 95% CI for the Kaplan-Meier estimates. Descriptive statistics will be used to evaluate the DOR achieved with the protocol therapy and with the most recent prior systemic therapy.
Overall survival (OS) (Phase I) | From the date of study entry up to 3 years
  OS will be estimated using Kaplan-Meier methodology. Greenwood's formula will be used to calculate 95% CI for the Kaplan-Meier estimates.
Progression-free survival (PFS) (Phase I) | From entry onto study up to 3 years
  PFS will be estimated using Kaplan-Meier methodology. Greenwood's formula will be used to calculate 95% CI for the Kaplan-Meier estimates.
ORR (Phase II) | Up to 10 years
  Assessed using Revised Response (Cheson) and Deauville criteria. The analysis of ORR between two arms will be performed using the CMH test stratifying on prior BV (yes vs. no) and age (< 18 vs. >= 18). Multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes.
PFS (or modified PFS) (Phase II) | From randomization up to 10 years
  PFS will be estimated using Kaplan-Meier methodology and compared between arms using stratified log-rank test. Greenwood's formula will be used to calculate 95% confidence intervals for the Kaplan-Meier estimates. Cox proportional regression model will be used to estimate hazard ratios (95% CI) and assess the relationship between other prognostic factors with time-to-event outcome. Point estimates of all endpoints will be accompanied by the corresponding 95% confidence intervals.
OS (Phase II) | From randomization up to 10 years
  OS will be estimated using Kaplan-Meier methodology and compared between arms using stratified log-rank test. Greenwood's formula will be used to calculate 95% confidence intervals for the Kaplan-Meier estimates. Cox proportional regression model will be used to estimate hazard ratios (95% CI) and assess the relationship between other prognostic factors with time-to-event outcome. Point estimates of all endpoints will be accompanied by the corresponding 95% confidence intervals.
DOR (Phase II) | From the documented beginning of response up to 10 years
  DOR, will be estimated using Kaplan-Meier methodology and compared between arms using stratified log-rank test. Greenwood's formula will be used to calculate 95% confidence intervals for the Kaplan-Meier estimates. Cox proportional regression model will be used to estimate hazard ratios (95% CI) and assess the relationship between other prognostic factors with time-to-event outcome. Point estimates of all endpoints will be accompanied by the corresponding 90% confidence intervals. The DOR achieved with the most recent prior systemic therapy will be collected on the case report forms, and descriptive statistics will be used to evaluate the DOR achieved with the protocol therapy and with the most recent prior systemic therapy.

OTHER OUTCOMES:
Change in the percentage of activated T cells and natural killer cells (Phase I and II) | Baseline (Time 1) to 9 weeks (Time 3, time of first re-staging)
  These quantities of interest will be calculated for each patient and the Wilcoxon signed-rank test will be used to test for significant difference between the time points. Using Wilcoxon rank sum test (two-sided type I error of 0.1), differences between those who progress or die within one year versus (vs.) those who are event-free at one year will be evaluated.
Change in the percentages of activated T cells and natural killer cells (Phase I and II) | Day 1 of cycle 2 (Time 2) or 9 weeks (Time 3) to up to 6 weeks after completion of study treatment (Time 4, end of study)
  These quantities of interest will be calculated for each patient and the Wilcoxon signed-rank test will be used to test for significant difference between the time points. Using the Wilcoxon rank sum test (two-sided type I error of 0.1), differences between those who progress or die within one year vs. those who are event-free at one year will be evaluated.
Effects of combinations on systemic immunity (Phase I and II) | Baseline to up to 6 weeks after completion of study treatment
Pre- and post-treatment levels of cytokines and T cell specific biomarkers (Phase I and II) | Baseline to up to 6 weeks after completion of study treatment
  Pre- and post-treatment levels of these markers will be compared using the Wilcoxon signed-rank test with two-sided type I error of 0.1. Marker levels between patients who fail at 1-year vs. patients who are event-free at 1-year will be evaluated. Given limited data, the analyses of PD-1, co-expression of Tim-3 with PD-1, ICOS, sCD30, galectin-1 and the peripheral blood absolute lymphocyte to monocyte ratio will be mainly exploratory and will be summarized descriptively at the time-points described above. The association with PFS will be explored.
Differentially expressed genes between two groups (patients who fail at 1-year vs. patients who are event-free at 1-year or responders vs. non-responders) (Phase I and II) | 1 year
  Assessed using gene expression profiling (GEP). Differentially expressed genes will be identified using a rank-based method developed by Dr. Hong (RankProd, R package, Bioconductor Project) with multiple comparison adjustment using a false discovery rate approach. A two-way unsupervised hierarchical clustering analysis will be applied to both the genes and the samples to illustrate whether GEP can separate two groups or is associated with other clinical factors. The genes ranked as most significant will be assessed by gene ontology and pathway analysis for their potential functions in lymphoma biology and treatment failure.
Microbiome analysis (Phase I and II) | Completion of study treatment
  Will compare the gut microbiome between Hodgkin lymphoma (HL) patients and healthy controls with respect to global diversity, taxonomic abundance, and bacterial functional pathways. The relative abundance of each taxon (phyla to genera) and functional pathways among different groups will be statistically compared in univariate analysis using t-test (or Wilcoxon test) and in multivariate analysis using logistic regression. Global diversity tests and multivariate analysis for taxonomic abundance and functional pathways will be adjusted for potential confounders (age, gender, race, and body mass index) in the comparisons of HL patients and controls, and further adjusted for stage and grade when examining the clinical response among HL patients.
Absolute maximum standard uptake value (SUVmax) (Phase II) | Up to cycle 10
  Image data will be evaluated using Lugano response criteria with various D 5PS cut-offs in the entire cohort and in different therapy cohorts to determine if the existing set of criteria is sufficient to segregate the group into various response categories. Will correlate PFS, event free survival (EFS), OS 5PS in two reading settings (1-3 [negative] vs 4-5 [positive] and D 5PS 1-4 [negative] vs 5 [positive]) (Kaplan-Meier [KM] curve and log-rank testing).
Metabolic whole body tumor volume (MTV) and tumor lesion glycolysis (TLG) | Up to cycle 10
  Image data will be evaluated using Lugano response criteria with various D 5PS cut-offs in the entire cohort and in different therapy cohorts to determine if the existing set of criteria is sufficient to segregate the group into various response categories. Will correlate PFS, EFS, OS 5PS in two reading settings (1-3 [negative] vs 4-5 [positive] and D 5PS 1-4 [negative] vs 5 [positive]) (KM curve and log-rank testing).
Percent change in SUVmax, MTV and TLG between baseline and during therapy | Baseline up to cycle 10
  Image data will be evaluated using Lugano response criteria with various D 5PS cut-offs in the entire cohort and in different therapy cohorts to determine if the existing set of criteria is sufficient to segregate the group into various response categories. Will correlate PFS, EFS, OS 5PS in two reading settings (1-3 [negative] vs 4-5 [positive] and D 5PS 1-4 [negative] vs 5 [positive]) (KM curve and log-rank testing).
Percent change in size (sum of perpendicular diameters [SPD]) on computed tomography (CT) | Baseline up to cycle 10
  Image data will be evaluated using Lugano response criteria with various D 5PS cut-offs in the entire cohort and in different therapy cohorts to determine if the existing set of criteria is sufficient to segregate the group into various response categories. Will correlate PFS, EFS, OS 5PS in two reading settings (1-3 [negative] vs 4-5 [positive] and D 5PS 1-4 [negative] vs 5 [positive]) (KM curve and log-rank testing).
Absolute CT tumor volumes | Up to cycle 10
  Image data will be evaluated using Lugano response criteria with various D 5PS cut-offs in the entire cohort and in different therapy cohorts to determine if the existing set of criteria is sufficient to segregate the group into various response categories. Will correlate PFS, EFS, OS 5PS in two reading settings (1-3 [negative] vs 4-5 [positive] and D 5PS 1-4 [negative] vs 5 [positive]) (KM curve and log-rank testing).
Percent change in CT size (SPD) and in CT tumor volume between baseline and during therapy | Baseline up to cycle 10
  Image data will be evaluated using Lugano response criteria with various D 5PS cut-offs in the entire cohort and in different therapy cohorts to determine if the existing set of criteria is sufficient to segregate the group into various response categories. Will correlate PFS, EFS, OS 5PS in two reading settings (1-3 [negative] vs 4-5 [positive] and D 5PS 1-4 [negative] vs 5 [positive]) (KM curve and log-rank testing).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine S Diefenbach, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (482):
- United States (482):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Mercy Health - Paducah Cancer Center, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Diefenbach C, Jegede O, Wang V, Ansell SM, Kostakoglu L, Steidl C, Natkunam Y, Scott DW, Ambinder RF, David KA, Advani RH, Bartlett NL, Robertson MJ, Thomas SP, Cohen JB, Ibrahimi S, Goyal G, Mehta-Shah N, Amengual JE, Forlenza CJ, Cole PD, Duan F, Kelly KM, Kahl BS. A Randomized Phase 2 Study of Ipilimumab, Nivolumab, and Brentuximab Vedotin in Patients with Relapsed Hodgkin Lymphoma. Blood. 2026 Feb 9:blood.2025029546. doi: 10.1182/blood.2025029546. Online ahead of print. PMID 41662628
- [Derived] Gonzalez-Kozlova E, Huang HH, Jagede OA, Tuballes K, Del Valle DM, Kelly G, Patel M, Xie H, Harris J, Argueta K, Nie K, Barcessat V, Moravec R, Altreuter J, Duose DY, Kahl BS, Ansell SM, Yu J, Cerami E, Lindsay JR, Wistuba II, Kim-Schulze S, Diefenbach CS, Gnjatic S. Tumor-Immune Signatures of Treatment Resistance to Brentuximab Vedotin with Ipilimumab and/or Nivolumab in Hodgkin Lymphoma. Cancer Res Commun. 2024 Jul 1;4(7):1726-1737. doi: 10.1158/2767-9764.CRC-24-0252. PMID 38934093
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794
- [Derived] Diefenbach CS, Hong F, Ambinder RF, Cohen JB, Robertson MJ, David KA, Advani RH, Fenske TS, Barta SK, Palmisiano ND, Svoboda J, Morgan DS, Karmali R, Sharon E, Streicher H, Kahl BS, Ansell SM. Ipilimumab, nivolumab, and brentuximab vedotin combination therapies in patients with relapsed or refractory Hodgkin lymphoma: phase 1 results of an open-label, multicentre, phase 1/2 trial. Lancet Haematol. 2020 Sep;7(9):e660-e670. doi: 10.1016/S2352-3026(20)30221-0. PMID 32853585